CLINICAL TRIAL: NCT06537687
Title: Relational Agents in Cervical Cancer Education (RACE)
Acronym: RACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radhika Gogoi (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Sponsor-Investigator, Radhika Gogoi, Principal Investigator, Associate Professor, Barbara Ann Karmanos Cancer Institute
Organization: Barbara Ann Karmanos Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-031
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Cervix Cancer; Human Papilloma Virus; Vaginal Cancer; Vulvar Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): The control group will be given a standardized handout
  Interventions: Other: Control
- Intervention (Experimental): The intervention group will be shown an educational video
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Control — A standardized handout on HPV and vaccine education will be given
  Arms: Control
Other: Intervention — A video about HPV and vaccines on a tablet provided by a research assistant
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to assess the feasibility of using interactive teaching to educate cervical cancer patients about Human papillomavirus (HPV) and HPV vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Patients with an ICD9 diagnosis of cervical/vaginal/vulvar cancer or dysplasia receiving care at Karmanos Cancer Institute or OU Health Stephenson Cancer Center

Exclusion Criteria:

* Patients who are recorded in the EHR as requesting to be removed from research
* Non-English speakers
* Any cognitive disability that prevents informed consent
* Any individual recruited in previous phases of the Study will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Participation Rate | Up to 6 weeks
  The Ratio of the number of participants to the number of patients asked to join the clinical trial
Survey Completion Rate | Up to 6 Weeks
  The Ratio of the number of participants who complete the survey to the number of participants overall.

SECONDARY OUTCOMES:
Change in intention to discuss HPV vaccination | Up to 6 weeks
  Changes from pre to post/follow up on intervention survey
Change in Health Literacy | Up to 6 weeks
  Changes in knowledge of HPV virus and prevention from pre to post/follow up survey
Change in social norms and behaviors | Up to 6 weeks
  Changes in social norms and behavioral control measures from pre and post/follow-up survey
Change in Stigma | Up to 6 weeks
  Changes in stigma measures in pre and post/follow up surveys

CONTACTS AND LOCATIONS:
Overall Officials: Radhika Gogoi, M.D. PhD, Principal Investigator — Karmanos Cancer Center
Locations (2):
- United States (2):
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT06537687/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT06537687/ICF_001.pdf